CLINICAL TRIAL: NCT06249035
Title: Feasibility of Transesophageal Echocardiography in Patients With Cardiac Arrest in Emergency Departments in the Netherlands
Brief Title: Feasibility of TEE During Cardiac Arrest in Dutch Emergency Departments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDTEE2024
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Arrest
Keywords: transoesophageal echocardiography; POCUS; Emergency Department
MeSH Terms: conditions — Heart Arrest; Emergencies | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Intervention Model Description: TEE will be performed on all patients that are eligible for inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEE as POCUS modality. (Experimental): TEE will be performed during cardiac arrest.
  Interventions: Diagnostic Test: Transoesophageal echocardiography (TEE)

INTERVENTIONS:
Diagnostic Test: Transoesophageal echocardiography (TEE) — TEE is a diagnostic modality in which an ultrasound probe is inserted via the oesophagus in order to visualize the heart.

SUMMARY:
The goal of this feasibility study is to learn if Dutch ED providers are able to use transesophageal echocardiography during cardiac arrest.

The main question it aims to answer is:

• are the ED providers able to determine the area of maximal compression of the heart using TEE

DETAILED DESCRIPTION:
Point-of-care ultrasound is a valuable diagnostic tool during cardiopulmonary resuscitation (CPR) in cardiac arrest and its use is recommended by international guidelines. Transthoracic echocardiography (TTE) is most commonly used, but has certain limitations. Image acquisition can be challenging due to patient specific factors such as body habitus. Also image quality may be impacted by the limited acquisition time during CPR pulse checks. Furthermore, observational data suggests that pulse checks are prolonged due to TTE, while minimizing interruption of chest compressions is emphasized for better CPR outcomes in the guidelines. Transesophageal ultrasound (TEE) is a possible alternative for TTE. It has the theoretical advantage of superior image quality and thereby possible reductions of chest compression delays. Furthermore, TEE gives the opportunity determine which part of the heart is compressed most effectively, which is referred to as the area of maximal compression (AMC). Animal studies showed that an AMC located over the left ventricle positively influenced hemodynamics and return of spontaneous circulation (ROSC) compared to an AMC over the aortic root. In human studies, data also suggests that AMC located on the left ventricle, as measured by TEE, may positively influence prognosis.

In the Netherlands, TEE is currently not used in emergency departments during cardiac arrest. The purpose of this study is to investigate if point-of-care TEE can be used effectively and safely by providers and teams that have not previously used this modality. Given the paramount importance of quality of chest compressions, the ability of the providers to assess the location of the AMC will be the main focus of this feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiac arrest > 18 year in the emergency department.

Exclusion Criteria:

* Patients with known upper gastro-intestinal malignancy or strictures, previous upper gastro-intestinal surgery or radiation, or known esophageal varices.
* Patient with a do-not-resuscitate order, pregnant patients and traumatic cardiac arrest.
* No trained TEE provider available.
* ROSC at arrival.
* Decision by the team to stop resuscitation at arrival at the emergency department due of prognosis.
* Other life saving interventions which are prioritized over TEE by the resuscitation team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Area of maximal compression (AMC) | First 30 minutes of cardiac arrest treatment in the ED.
  The percentage of patients in which providers are able to determine the location of the AMC during cardiac arrest.

SECONDARY OUTCOMES:
Location of AMC | First 30 minutes of cardiac arrest treatment in the ED.
  The echographic location of the AMC, subcategorised as: left ventricle, left ventricular outflow tract/aortic root, other, not able to determine AMC
Accuracy of AMC | First 30 minutes of cardiac arrest treatment in the ED.
  Accuracy of AMC defined as correlation between providers interpretation of AMC and reviewers interpretation of AMC
Safety of TEE | First 30 minutes of cardiac arrest treatment in the ED.
  Incidence of complications of TEE
Intubation | First 30 minutes of cardiac arrest treatment in the ED.
  Need for intubation for using TEE and duration of intubation
Time to image | First 30 minutes of cardiac arrest treatment in the ED.
  Time from start ED treatment to first TEE image

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No